CLINICAL TRIAL: NCT03747003
Title: Gonadal Function in Young to Middle Aged HIV-infected Men Assessed by Isotopic Dilution-liquid Chromatography-mass Spectrometry (ID-LC-MS/MS) and Chemiluminescent Immunoassay
Brief Title: Gonadal Function in Young to Middle Aged HIV-infected Men
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, Associate Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 15/13
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Human Immunodeficiency Virus; Hypogonadism, Male; Erectile Dysfunction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Eunuchism; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for hormonal assay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-infected male patients: Male patients (age 18-50 years) with HIV-infection and ongoing HAART therapy No intervention is provided
  Interventions: Other: No intervention is provided

INTERVENTIONS:
Other: No intervention is provided — No intervention is provided

SUMMARY:
HIV infection is associated to premature decline of serum testosterone. However, prevalence and biochemical characterization of hypogonadism in HIV-infected men are still to be well defined. HIV-infection is strongly associated to erectile dysfunction in men, but preliminary data suggest that it is poorly associated with serum testosterone in this context.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the gonadal function of young to middle aged HIV-infected men in order to characterize hypogonadism by assessing circulating total testosterone with either Liquid Chromatography tandem Mass Spectrometry (LC-MS/MS) or chemiluminescent immunoassay. Furthermore, secondary aim is to assess the erectile function through the use of validated questionnaires (International Index of Erectile Function (IIEF) 15 and 5).

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age 18-50 years
* HIV-infection
* Ongoing Highly Active Antiretroviral Therapy

Exclusion Criteria:

* Previous treatment with androgens, anti-androgens
* Severe liver insufficiency
* Severe renal insufficiency

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Cohort of Young-to-Middle Aged HIV-infected Patients
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Serum total testosterone | Assessed only once at the moment of enrollment with liquid chromatography tandem mass spectrometry
  From blood sample - unit of measurement ng/dL
Serum total testosterone | Assessed only once at the moment of enrollment with chemiluminiscent immunoassay
  From blood sample - unit of measurement ng/dL

SECONDARY OUTCOMES:
Serum free testosterone | Calculated only once at the moment of enrollment
  Calculated formula (Vermeulen equation)
Score at IIEF questionnaire | Assessed only once at the moment of enrollment
  Total score at erectile function domain of IIEF-15 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero - Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No